CLINICAL TRIAL: NCT06431750
Title: Prospective Observational Study to Evaluate Secukinumab Treatment Effectiveness in Pediatric Patients With Active Juvenile Enthesitis-related or Psoriatic Arthritis (Toddler)
Brief Title: Prospective Observational Study to Evaluate Secukinumab Treatment Effectiveness in Pediatric Patients With Active Juvenile Enthesitis-related or Psoriatic Arthritis
Acronym: Toddler
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457FRU02
Record Dates: First submitted 2024-04-30; First posted 2024-05-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile Idiopathic Arthritis; JIA; Secukinumab; Cosentyx
MeSH Terms: conditions — Arthritis, Juvenile | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Secukinumab: pediatric patients with active ERA/jPsA for whom routine treatment with secukinumab according to the approved national label is initiated during 4 to 8 weeks prior to enrollment
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — This is an observational study, there is no treatment allocation.

SUMMARY:
This is a multicenter, non-interventional, cohort study in pediatric patients with active juvenile enthesitis-related or psoriatic arthritis

DETAILED DESCRIPTION:
Rheumatologists and pediatricians actively managing pediatric Enthesitis-related Arthritis (ERA) and Juvenile Psoriatic Arthritis (jPsA) in different regions of Russia are planned to participate in the study. To be include in this study, physicians must consult more than 10 pediatric patients with ERA/jPsA in a typical month. Any pediatric patients with active ERA/jPsA who started secukinumab treatment (index date) within 4-8 weeks prior to inclusion can be enrolled. At the inclusion retrospective data collection is planned, then data will be collected 3 months of treatment), 6, 12, 18, and 24 months after index date. Therefore, maximum duration of prospective observation is expected to be 23 months. Data collection schedule fits routine (Juvenile Idiopathic Arthritis) JIA management guidelines for patients receiving biologics stating that treatment effectiveness should be evaluated at 3 and 6 months after biologic initiation and every 6 months thereafter. At each visit effectiveness and tolerability parameters, as well as the patients' Quality of life (QoL) will be documented. Retrospective data will be collected for medical history and JIA treatment, including secukinumab before inclusion, as well to describe all necessary parameters since the Index date. Expected look-back period is 12 months.

Initiation of secukinumab treatment will be considered the index date.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and legal representative's permission for study participation obtained prior to beginning of participation in the study.
2. Age ≥6 to <18 years old.
3. Recognized physician diagnosis of active ERA or jPsA:

   * ERA per ILAR criteria:

     * Peripheral arthritis and enthesitis, or
     * Arthritis or enthesitis, plus ≥ 3 months of inflammatory back pain and sacroiliitis on imaging, or
     * Arthritis or enthesitis plus 2 of the following: sacroiliac joint tenderness; inflammatory back pain; presence of HLA-B27 antigen; acute (symptomatic) anterior uveitis; and history of a spondyloarthritis in a first-degree relative.
   * jPsA per ILAR criteria

     * Arthritis and psoriasis, or
     * arthritis and at least 2 of the following:

       * Dactylitis
       * Nail pitting or onycholysis
       * Psoriasis in a first-degree relative.
4. Patient was prescribed with secukinumab within 4-8 weeks before inclusion.
5. Decision for secukinumab prescription was made by the attending physician according to the approved national label during routine clinical practice, regardless of this non-interventional study conduct.
6. The Purified Protein Derivative (PPD) Skin Test for Tuberculosis and/or Negative T-SPOT test and/or TB-feron test before secukinumab treatment and every 6 months.

Exclusion Criteria:

1. Known or suspected severe hypersensitivity for secukinumab, formulation excipients, or injection device components (i.e., latex).
2. Chronic recurrent infections.
3. Clinically significant infection exacerbation, including active tuberculosis.
4. Age <6 years or ≥18 years.
5. Pregnancy and breastfeeding.
6. Patients participating in parallel in an interventional clinical trial.
7. Patients participating in parallel in other Novartis-sponsored non-interventional study generating primary data for secukinumab.
8. Patients within the safety follow-up phase of interventional study.
9. Active inflammatory bowel disease at inclusion.
10. Patients who received any vaccine within 4 weeks prior to secukinumab initiation.
11. Any medical or psychological condition in the investigator's opinion which may prevent the study participation.
12. Concomitant conditions (Candida infections, other infections, inflammatory bowel disease [IBD], uveitis, skin and nail psoriasis for ERA patients, hepatitis B, hepatitis C, tuberculosis).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with active ERA/jPsA for whom routine treatment with secukinumab according to the approved national label is initiated during 4 to 8 weeks prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Drug survival rate | 24 months
  Drug survival is defined as time from the index date (defined as secukinumab treatment initiation) until discontinuation of secukinumab
American College of Rheumatology pediatric (ACR Pedi) 30/50/70/90 achievement rates | Month 3, Month 6, Month 12, Month 18, and Month 24
  The ACR Pedi 30/50/70/90 is defined as a minimum of 30/50/70/90 percent improvement from baseline in a minimum of 3 out of 6 components, with no more than 1 component worsening by >30/50/70/90 percent.
  The ACR Pedi consists of 6 core criteria:
  1. physician global assessment (PGA) of disease activity (visual analog scale [VAS]) where 0 represents no disease activity and 100 represents the most disease activity
  2. assessment of overall well-being (VAS) where 0 represents very well and 100 represents very poor for overall well-being
  3. functional ability (assessed using the Childhood Health Assessment Questionnaire [CHAQ]);
  4. number of joints with active arthritis (defined as joints with swelling not caused by deformity or joints, in the absence of swelling, with limitation of passive motion accompanied by pain, tenderness, or both)
  5. number of joints with limited range of motion
  6. laboratory marker of inflammation (C-reactive protein [CRP]).
Clinical remission/inactive disease rates by Wallace criteria | Month 3, Month 6, Month 12, Month 18, and Month 24
  To state the absence of disease activity (inactive phase of the disease), the patient must meet all of the listed criteria.
  * absence of joints with active arthritis,
  * absence of fever, rash, serositis, splenomegaly or generalized lymphadenopathy typical of juvenile arthritis;
  * absence of active uveitis,
  * normal ESR and (or) CRP,
  * absence of disease activity according to the doctor's general assessment (VAS),
  * morning stiffness less than 15 minutes.

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnaire (CHAQ) score | Up to 24 months
  Describes the child's usual activities in eight domains over the past week. It include dressing, getting up, eating, walking, hygiene, reaching overhead objects, grip and activities. Each question is scored from 0 to 3 (0 = no difficulty, 1 = some difficulty, 2 = much difficulty and 3 = unable to do). The score for each of the eight functional areas will be averaged to calculate the disability index.
Physician global assessment of disease activity | Up to 24 months
  Physician global assessment of disease activity assessed on a VAS scale of 0 [no activity] to 10 [extreme activity]
Patient/legal representative global assessment of disease activity | Up to 24 months
  Patient/legal representative global assessment of disease activity assessed on a VAS scale of 0 [no activity] to 10 [extreme activity]
Time to treatment failure | Up to 24 months
  Time to treatment failure defined as time from index date to loss of ACR Pedi 30, 50, and 70 response.
Proportion of patients not achieving ACR Pedi 30 response | Month 3
  The ACR Pedi 30 is defined as a minimum of 30 percent improvement from baseline in a minimum of 3 out of 6 components, with no more than 1 component worsening by >30 percent.
  The ACR Pedi consists of 6 core criteria:
  1. physician global assessment (PGA) of disease activity (visual analog scale [VAS]) where 0 represents no disease activity and 100 represents the most disease activity
  2. assessment of overall well-being (VAS) where 0 represents very well and 100 represents very poor for overall well-being
  3. functional ability (assessed using the Childhood Health Assessment Questionnaire [CHAQ]);
  4. number of joints with active arthritis (defined as joints with swelling not caused by deformity or joints, in the absence of swelling, with limitation of passive motion accompanied by pain, tenderness, or both)
  5. number of joints with limited range of motion
  6. laboratory marker of inflammation (C-reactive protein [CRP]).
Disease activity index in 71 joints Juvenile Arthritis Disease Activity Score (JADAS71) | Up to 24 months
  Score to evaluate the number of joints inflamed. A joint is considered to be inflamed when at leats two of the following criteria are present:
  * pain
  * Swelling
  * limited motion. The score range (total) is from 0-101, where higher scores indicate worse outcome.
Juvenile Spondyloarthritis (JSpA) Disease Activity - JSpADA | Up to 24 months
  The JSpADA score is a comprehensive
  clinical assessment tool designed to measure the impact of juvenile spondyloarthritis on the patient. The JSpADA scale includes 8 indicators that assess the signs and symptoms of spondyloarthritis. Patients receive an overall score based on scores on each of 8 indicators. There are two options for assessing morning stiffness, clinical sacroiliitis, uveitis and back mobility: presence or absence. Number of joints with active arthritis: 0 joints = 0; 1-2 joints = 0.5; > 2 joints = 1; Number of active enthesites: 0 = 0; 1-2 = 0.5; > 2 = 1; Patient-Reported Pain Score (VAS 0-10): 0 = 0; 1-4 = 0.5; 5-10 = 1; Assessment of ESR or CRP level: normal = 0; 1-2x = 0.5; > 2x = 1.
  As a result, we add up the scores for the obtained indicators and get an overall score, and the higher it is, the higher the disease activity.
Psoriasis Area and Severity Index (PASI) for patients with Juvenile Psoriatic Arthritis (jPsA) | Up to 24 months
  Psoriasis Area and Severity Index (PASI) for patients with Juvenile Psoriatic Arthritis (jPsA) to be provided. Score can range from 0 (no disease) to 72 (maximal disease).
Number of participants by reasons of secukinumab discontinuation | Up to 24 months
  Reasons for discontinuation:
  * lack of efficacy,
  * adverse events
  * administrative reasons (no medication available in the hospital, etc.)
  * lack of patient's adherence
  * patient's or legal representative's wish
  * other.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No